CLINICAL TRIAL: NCT01016470
Title: Efficacy of Nutritional Supplement VIUSID/ALZER in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAT-0916-CU
Record Dates: First submitted 2009-09-28; First posted 2009-11-19 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Viusid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- A (Experimental): VIUSID/ALZER. The purpose of the study is to evaluate whether Viusid/Alzer Nutritional supplements, could improve the progression disease, in patients with early PD by UPDRS motor
  Interventions: Dietary Supplement: VIUSID/ALZER

INTERVENTIONS:
Dietary Supplement: VIUSID/ALZER — VIUSID/ALZER, 3 per day, oral, one year
  Arms: A
Dietary Supplement: Placebo — Placebo Viusid and Placebo Alzer, 3 per day, oral, one year
  Arms: B

SUMMARY:
The purpose of the study is to evaluate whether Viusid/Alzer Nutritional supplements, could improve the progression disease, in patients with Parkinson's Disease (PD).

DETAILED DESCRIPTION:
Periodical measures of the clinical features with UPDRS will be done at the beginning, each three months until two years. Each group will be compare to evaluate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical of PD, with the criteria of Brain Bank of London with early stage.
* Informed consent.

Exclusion Criteria:

* Presence of another disease not well controlled.
* Patient with atypical features.
* Patient with advanced Parkinson's disease.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Periodical measures of the clinical features with Unified Parkinson Disease Rating Scale (UPDRS) will be done at the beginning, every three months until one year (end of the treatment) | one year

SECONDARY OUTCOMES:
Hoehn-Yarh will be done at the beginning, every three months until one year (end of the treatment) | one year
Dosage levodopa will be done at the beginning, every three months until one year (end of the treatment) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Guiroud, PhD, Principal Investigator — "Salvador Allende" Hospital
Locations (1):
- "Salvador Allende Hospital", Havana, La Habana, Cuba

REFERENCES:
- See also: Related Info — http://www.catalysis.es